CLINICAL TRIAL: NCT02355223
Title: Finding and Treating Unsuspected and Resistant TB to Reduce Hospital Transmission
Acronym: FAST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Hospital Nacional Hipólito Unanue (Unknown); Socios En Salud Sucursal, Peru (Other); Hospital Nacional Arzobispo Loayza (Other); Hospital Nacional Sergio Bernales (Unknown)
Responsible Party: Principal Investigator, Edward Anthony Nardell, MD, Associate Physician, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2014P002396
Record Dates: First submitted 2015-01-28; First posted 2015-02-04 (Estimated); Last update posted 2018-01-12 (Actual); Status verified 2018-01

CONDITIONS: Tuberculosis
Keywords: Tuberculosis; Infection Control; Transmission
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FAST Implementation (Other): This single center study will consist of introducing a TB screening program called FAST (Find cases Actively, Separate safely, and Treat Effectively) within the hospital among patients presenting for care who have cough or TB risk factors, and testing them for tuberculosis using a combination of rapid screening and diagnostics tools. The study will evaluate the process of implementation as well as the impact on reducing tuberculosis transmission to health care workers over successive years.
  Interventions: Other: FAST

INTERVENTIONS:
Other: FAST — See information in arm description

SUMMARY:
The study is designed to evaluate the clinical impact of a novel strategy for tuberculosis (TB) infection control known as FAST (Find cases Actively based on cough surveillance, Separate temporarily, and Treat effectively). It is anticipated that this will decrease time to effective treatment initiation and also decrease transmission of TB to health care workers.

DETAILED DESCRIPTION:
There is longstanding evidence that tuberculosis (TB) transmission is not from TB patients on effective treatment, but from unsuspected cases, and cases with unsuspected drug resistance. This study seeks to investigate the implementation of a refocused TB transmission control approach that we call FAST (Find cases Actively based on cough surveillance, Separate temporarily, and Treat effectively based on molecular drug-susceptibility testing [DST]). We will conduct this study at Hospital Nacional Hipólito Unanue in Lima, Peru. Our hypothesis is that FAST will reduce delays in identifying infectious TB patients (and unsuspected drug resistance) entering the hospital, facilitate timely effective therapy, and thereby reduce the risk of TB transmission in a cost-effective manner. We will assess the impact of FAST on TB transmission by evaluating IGRA conversions among health care workers at the intervention site, Hospital Nacional Hipolito Unanue (HNHU), and two control sites, Hosptial Nacional Arzobispo Loayza (HNAL) and Hospital Nacional Sergio Bernales (HNSB). We will also evaluate acceptability and barriers to/facilitators of FAST, novel screening strategies, and health care worker IGRA testing using a mixed methods approach.

ELIGIBILITY:
Inclusion Criteria (for patients):

* adult (≥ 18 years) patients who are receiving care in the emergency department or being admitted for inpatient care from any other hospital area
* patient presenting with cough or TB risk factors of prior or current TB diagnosis and/or contact of an individual with TB
* able to participate by providing a sputum sample and/or exhaled breath test sample

Exclusion Criteria (for patients):

* no specific exclusion criteria at initial screening if the patient meets the above inclusion criteria.

Inclusion Criteria (for health care workers):

* being an employee or intern at Hospital Nacional Hipolito Unanue (HNHU), Hospital Nacional Arzobispo Loayza (HNAL) or Hospital Nacional Sergio Bernales (HNSB) and deemed to be at risk of exposure to tuberculosis based on line of work
* age ≥ 18 years
* willing and able to provide informed consent for participation

Exclusion Criteria (for health care workers):

* no specific exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11060 (Estimated)
Dates: Start 2016-08; Primary Completion 2020-02 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Reduction of time to TB diagnosis and treatment for patients and TB infection rates in health care workers. | 5 years
  Time to diagnosis and Time to effective treatment initiation

SECONDARY OUTCOMES:
Sensitivity and specificity of a novel exhaled breath test (EBT) and digital chest X-ray with computer assisted detection (dCXR/CAD4TB) as "rule-out" screening tests for tuberculosis in coughing patients | 5 years
  Sensitivity and specificity of EBT and dCXR/CAD4TB will be calculated along with negative predictive value
Costs and cost-effectiveness of FAST | 5 years
  Cost effectiveness analysis
Acceptability of FAST, novel screening strategies, and health care worker testing for latent tuberculosis. | 5 years
  Qualitative data collection using surveys and focus groups to assess acceptability and barriers

CONTACTS AND LOCATIONS:
Overall Officials: Edward Nardell, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Hospital Nacional Hipolito Unanue, Lima, Peru

REFERENCES:
- [Background] Joshi R, Reingold AL, Menzies D, Pai M. Tuberculosis among health-care workers in low- and middle-income countries: a systematic review. PLoS Med. 2006 Dec;3(12):e494. doi: 10.1371/journal.pmed.0030494. PMID 17194191
- [Background] Brennen C, Muder RR, Muraca PW. Occult endemic tuberculosis in a chronic care facility. Infect Control Hosp Epidemiol. 1988 Dec;9(12):548-52. doi: 10.1086/645774. PMID 3235808
- [Background] Kantor HS, Poblete R, Pusateri SL. Nosocomial transmission of tuberculosis from unsuspected disease. Am J Med. 1988 May;84(5):833-8. doi: 10.1016/0002-9343(88)90060-5. PMID 3364442
- [Background] Moran GJ, McCabe F, Morgan MT, Talan DA. Delayed recognition and infection control for tuberculosis patients in the emergency department. Ann Emerg Med. 1995 Sep;26(3):290-5. doi: 10.1016/s0196-0644(95)70074-9. PMID 7661416
- [Background] Willingham FF, Schmitz TL, Contreras M, Kalangi SE, Vivar AM, Caviedes L, Schiantarelli E, Neumann PM, Bern C, Gilman RH; Working Group on TB in Peru. Hospital control and multidrug-resistant pulmonary tuberculosis in female patients, Lima, Peru. Emerg Infect Dis. 2001 Jan-Feb;7(1):123-7. doi: 10.3201/eid0701.010117. PMID 11266302
- [Background] Bonifacio N, Saito M, Gilman RH, Leung F, Cordova Chavez N, Chacaltana Huarcaya J, Vera Quispe C. High risk for tuberculosis in hospital physicians, Peru. Emerg Infect Dis. 2002 Jul;8(7):747-8. doi: 10.3201/eid0807.010506. No abstract available. PMID 12095450
- [Background] ANDREWS RH, DEVADATTA S, FOX W, RADHAKRISHNA S, RAMAKRISHNAN CV, VELU S. Prevalence of tuberculosis among close family contacts of tuberculous patients in South India, and influence of segregation of the patient on early attack rate. Bull World Health Organ. 1960;23(4-5):463-510. PMID 13683486
- [Background] Kamat SR, Dawson JJ, Devadatta S, Fox W, Janardhanam B, Radhakrishna S, Ramakrishnan CV, Somasundaram PR, Stott H, Velu S. A controlled study of the influence of segregation of tuberculous patients for one year on the attack rate of tuberculosis in a 5-year period in close family contacts in South India. Bull World Health Organ. 1966;34(4):517-32. PMID 5296379
- [Background] Rouillon A, Perdrizet S, Parrot R. Transmission of tubercle bacilli: The effects of chemotherapy. Tubercle. 1976 Dec;57(4):275-99. doi: 10.1016/s0041-3879(76)80006-2. PMID 827837
- [Background] Dharmadhikari AS, Mphahlele M, Venter K, Stoltz A, Mathebula R, Masotla T, van der Walt M, Pagano M, Jensen P, Nardell E. Rapid impact of effective treatment on transmission of multidrug-resistant tuberculosis. Int J Tuberc Lung Dis. 2014 Sep;18(9):1019-25. doi: 10.5588/ijtld.13.0834. PMID 25189547